CLINICAL TRIAL: NCT00660075
Title: A Randomized, Double-Blind, Placebo-Controlled, Crossover Study To Evaluate The Effects of Sitagliptin on Postprandial Plasma Lipoprotein Concentrations in Men With Type 2 Diabetes
Brief Title: Effects of Sitagliptin on Postprandial Lipemia in Men With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Patrick Couture, Médecin, Laval University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SITA001
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Results first posted 2012-12-11 (Estimated); Last update posted 2012-12-11 (Estimated); Status verified 2012-11

CONDITIONS: Diabetes Mellitus; Postprandial Lipemia
Keywords: Diabetes mellitus; Postprandial; Hyperlipidemia; Atherosclerosis
MeSH Terms: conditions — Diabetes Mellitus; Hyperlipidemias; Atherosclerosis | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Sitagliptin 100 mg/d for 6 weeks
  Interventions: Drug: Sitagliptin
- 2 (Placebo Comparator): Placebo for 6 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg/d for 6 weeks
  Arms: 1
Drug: Placebo — Placebo for 6 weeks
  Arms: 2

SUMMARY:
Sitagliptin is a potent and selective inhibitor of dipeptidyl peptidase IV (DPP-4), and has been shown to reduce fasting and postprandial glucose levels in patients with type 2 diabetes mainly through incretin hormone-mediated improvements in islet function. Although clinical studies to date indicate that fasting lipid levels are minimally affected by DPP-4 inhibitor treatment, animal studies suggested that DPP-4 inhibition reduce intestinal triglyceride (TG) absorption and apolipoprotein production and increased chylomicron catabolism. Therefore, the present study was designed to examine the effects of sitagliptin on postprandial lipemia in patients with type 2 diabetes. A possible reduction in postprandial atherogenic triglyceride-rich lipoproteins (TRL) levels by sitagliptin would add to therapeutic utility of this DPP-4 inhibitor and suggest the potential to reduce cardiovascular risk in patients with type 2 diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes as defined by the American Diabetes Association;
* Non-smoker;
* Body mass index between 25.0 and 40.0 kg/m2;
* Baseline HbA1c between 6.5 and 8.5%;
* Baseline fasting plasma glucose < 15.0 mmol/L;
* Plasma triglyceride levels between 1.5 and 8.0 mmol/L (135 and 710 mg/dl) at week and -4;
* Patients having received stable doses of metformin for at least 3 months before randomization;
* Subjects must be willing to give written informed consent and able to adhere to dosing schedule, visit schedule and phone follow-up assessment;
* Patients should be otherwise generally healthy, without elevations in hepatic transaminases or abnormal renal function or coagulation;
* Patients having normal TSH at screening.

Exclusion Criteria:

* Patients with extreme dyslipidemias, such as familial hypercholesterolemia will be excluded;
* Patients with type 1 diabetes, secondary form of diabetes or acute metabolic diabetic complications will be excluded;
* Patients having received or being treated with insulin or a thiazolidinedione within the past 6 months will be excluded;
* Subjects will be excluded if they have cardiovascular disease (CVD) (coronary heart disease, cerebrovascular disease or peripheral arterial disease) or if they are taking other medications known to affect lipoprotein metabolism (e.g. steroids, beta blockers, thiazide diuretics, lipid lowering agents, significant alcohol intake etc.);
* Subjects who are in a situation or have any condition that, in the opinion of the investigator, may interfere with optimal participation in the study;
* Individuals with a history of mental instability, drug or alcohol abuse or individuals who have been treated or are being treated for severe psychiatric illness that, in the opinion of the investigator, may interfere with optimal participation in the study;
* History of alcohol or drug abuse within the past 2 years. Patients must not take alcohol during the study;
* Disorders of the hematologic, digestive, or central nervous systems, including cerebrovascular disease and degenerative disease, that would limit study evaluation or participation;
* Known impairment of renal function (serum creatinine levels > 1.7 mg/dL for men), dysproteinemia, nephrotic syndrome, or other renal disease (24-hour urinary protein ≥3 ± 1 g);
* Active or chronic hepatobiliary or hepatic disease. In addition, patients with AST or ALT >2 x upper limit of the laboratory reference range will be excluded;
* Subjects with coagulopathy (prothrombin time [PT] or partial thromboplastin time [PTT] at Visit 1 >1.5 times control;
* Patients who are known to have tested positive for human immunodeficiency virus (HIV);
* Patients who are currently enrolled in another clinical study;
* Patients who have used any investigational drug within 30 days of the first clinic visit;
* Congestive heart failure NYHA Class III or IV. Uncontrolled cardiac arrhythmias within 3 months of study entry;
* Uncontrolled diabetes mellitus (HbA1c>8.5%) or other endocrine or metabolic disease known to influence serum lipids or lipoproteins. Clinically euthyroid subjects on replacement doses of thyroid hormone are eligible for enrollment.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Couture, MD, PhD, Principal Investigator — Laval University
Locations (1):
- Laval University Medical Center, Québec, Quebec, Canada

REFERENCES:
- [Derived] Tremblay AJ, Lamarche B, Deacon CF, Weisnagel SJ, Couture P. Effects of sitagliptin therapy on markers of low-grade inflammation and cell adhesion molecules in patients with type 2 diabetes. Metabolism. 2014 Sep;63(9):1141-8. doi: 10.1016/j.metabol.2014.06.004. Epub 2014 Jun 14. PMID 25034387

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Location: CHUL Medical Centre Date: Fall 2007, Winter 2008, Fall 2008
Pre-assignment Details: 2-weeks run-in period. 6-weeks treatment with sitagliptin 100mg/d or placebo. 4-weeks washout period. 6-weeks treatment with sitagliptin or placebo.
Groups:
- Placebo First, Then Sitagliptin: Participants were first administered placebo for 6 weeks followed by a washout period of 4 weeks and were then switched over to Sitagliptin 100 mg/d for 6 weeks.
- Sitagliptin First, Then Placebo: Participants were first administered Sitagliptin 100 mg/d for 6 weeks followed by a washout period of 4 weeks and were then switched over to placebo for 6 weeks.
Period: First Intervention (Week 1 to Week 6)
Arm/Group | Placebo First, Then Sitagliptin | Sitagliptin First, Then Placebo
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Washout Period (Week 7 to Week 10)
Arm/Group | Placebo First, Then Sitagliptin | Sitagliptin First, Then Placebo
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0
Period: Second Intervention (Week 11 to Week 16
Arm/Group | Placebo First, Then Sitagliptin | Sitagliptin First, Then Placebo
Started | 18 | 18
Completed | 18 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 18 | 18 | 36
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 16 | 32
  >=65 years | 2 | 2 | 4
Age Continuous [Mean (Standard Deviation); unit: years] | 57.4 (6.5) | 58.8 (6.3) | 58.1 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 6 | 6
  Male | 18 | 12 | 30
Region of Enrollment [Number; unit: participants]
  Canada | 18 | 18 | 36

OUTCOME MEASURES:

1. Primary Outcome: Measurement of the Area Under the Curve of Plasma Triglycerides (TG) Levels During Postprandial Period (Time 0,2,4,6,8 Hours)
Time Frame: At the end of the two 6-week interventions
Population: We analyzed all the subjects involved in the study. The analysis was per protocol. We compared data from the placebo phase with the sitagliptin phase.
Measure: Mean (Standard Deviation); unit: mmol*h/L
Groups:
- Sitagliptin 100 mg/d: Sitagliptin 100 mg/d for 6 weeks
Arm/Group | Placebo | Sitagliptin 100 mg/d
Number analyzed (Participants) | 36 | 36
mmol*h/L | 30.0 (14.5) | 27.1 (13.0)

ADVERSE EVENTS:
Arm/Group | Sitagliptin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 0/18 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No